CLINICAL TRIAL: NCT04003857
Title: Follow-up Study of Safety and Efficacy in Subjects Who Completed PNEUMOSTEM® Phase II (MP-CR-012) Clinical Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-CR-012-F/U
Record Dates: First submitted 2019-06-19; First posted 2019-07-01 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Bronchopulmonary Dysplasia; BPD
Keywords: Human Umbilical Cord Blood Derived Mesenchymal Stem Cells; Bronchopulmonary dysplasia; Premature infants
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PNEUMOSTEM® (Experimental): A single intratracheal administration of Pneumostem® (10.0 x 10^6 cells/kg)
  Interventions: Biological: PNEUMOSTEM®
- normal saline (Placebo Comparator): A single intratracheal administration of normal saline
  Interventions: Biological: normal saline

INTERVENTIONS:
Biological: PNEUMOSTEM® — A single intratracheal administration of PNEUMOSTEM® (1.0 x 10^7 cells/kg)
  Other Names: Human umbilical cord blood-derived mesenchymal stem cells
  Arms: PNEUMOSTEM®
Biological: normal saline — A single intratracheal administration of normal saline
  Arms: normal saline

SUMMARY:
This is a follow-up study to investigate the long-term safety and efficacy of PNEUMOSTEM® versus placebo, for the treatment of BPD in premature infants. Subjects who participated in and completed the initial stage of the Phase II trial (NCT03392467) will be followed-up until 60 months of corrected age

DETAILED DESCRIPTION:
Subjects who completed the initial stage of the Phase II clinical trial will be followed-up at 7 additional visits: 6, 12,18, 24 months corrected age, 36, 48, and 60 months after birth.

ELIGIBILITY:
Inclusion Criteria:

* Subject who enrolled in phase 2 clinical trial of PNEUMOSTEM® to evaluate efficacy and safety, and were administered with investigational product
* Subject with a written consent form signed by a legal representative or a parent upon explanation of the clinical trial

Exclusion Criteria:

* Subject whose parent or legal representative does not agree to participate in the study
* Subject who is considered inappropriate to participate in the study by the investigator

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory outcome: Number of hospitalizations | 6 months corrected age
  Total number of hospitalizations and the number of hospital stay due to respiratory infection
Respiratory outcome: Number of hospitalizations | 12 months corrected age
  Total number of hospitalizations and the number of hospital stay due to respiratory infection
Respiratory outcome: Number of hospitalizations | 18 months corrected age
  Total number of hospitalizations and the number of hospital stay due to respiratory infection is recorded and compared with control group
Respiratory outcome: Number of hospitalizations | 24 months corrected age
  Total number of hospitalizations and the number of hospital stay due to respiratory infection
Respiratory outcome: Number of hospitalizations | 36 months after birth
  Total number of hospitalizations and the number of hospital stay due to respiratory infection
Respiratory outcome: Number of hospitalizations | 39 months after birth
  Total number of hospitalizations and the number of hospital stay due to respiratory infection
Respiratory outcome: Number of hospitalizations | 42 months after birth
  Total number of hospitalizations and the number of hospital stay due to respiratory infection
Respiratory outcome: Number of hospitalizations | 45 months after birth
  Total number of hospitalizations and the number of hospital stay due to respiratory infection
Respiratory outcome: Number of hospitalizations | 48 months after birth
  Total number of hospitalizations and the number of hospital stay due to respiratory infection
Respiratory outcome: Number of hospitalizations | 51 months after birth
  Total number of hospitalizations and the number of hospital stay due to respiratory infection
Respiratory outcome: Number of hospitalizations | 54 months after birth
  Total number of hospitalizations and the number of hospital stay due to respiratory infection
Respiratory outcome: Number of hospitalizations | 57 months after birth
  Total number of hospitalizations and the number of hospital stay due to respiratory infection
Respiratory outcome: Number of hospitalizations | 60 months after birth
  Total number of hospitalizations and the number of hospital stay due to respiratory infection

SECONDARY OUTCOMES:
Mortality | 6, 12, 18, 24 months corrected age, 36, 48, and 60 months after birth
  check whether patient is alive or dead at evaluation time point
Growth measured by Z-score | 6, 12, 18, 24 months corrected age, 36, 48, and 60 months after birth
  Growth measured by Z-score
Neurological developmental status: Korean Developmental Screening Test for infants and children(K-DST) | 6, 12, 18, 24 months corrected age,36, 48, and 60 months after birth
  Neurological developmental status on Korean Developmental Screening Test for infants and children(K-DST)
Deafness or Blindness | 24 months corrected age
  Deafness: audiometry /Blindness: examination of extraocular muscle, fundus photography, optical biometry
Bayley Scales of Infant and Toddler Development (Third Edition) | 18~24months corrected age, 36~42months after birth
  Scale: cognitive, motor, language, social-emotional, adaptive behavior
Gross Motor Function Classification System for Cerebral Palsy | 24 months corrected age
  Gross Motor Function Classification System for Cerebral Palsy
Number of adverse events | 6, 12, 18, 24 months corrected age,36, 48, and 60 months after birth
  Number of adverse events
Number of admissions to Emergency Room (ER) | 6, 12, 18, 24months corrected age, 36, 39, 42, 45, 48, 51, 54, 57 and 60 months after birth
  Total number of admissions to Emergency Room (ER) and number of admission to Emergency Room (ER) due to respiratory infection at each evaluation time point
Medical treatment records | 6, 12, 18, 24months corrected age, 36, 39, 42, 45, 48, 51, 54, 57 and 60 months after birth
  whether or not, the patient is receiving medical treatment(use of oxygen, steroid, or bronchodilator, diuretics, Sildenafil) and if receiving treatment, the duration of the treatment at each evaluation time point

CONTACTS AND LOCATIONS:
Overall Officials: Wonsoon Park, MD, PhD, Principal Investigator — Department of Pediatrics, Samsung Medical Center; Ai-Rhan Kim, MD, PhD, Principal Investigator — Department of Neonatology, Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No